CLINICAL TRIAL: NCT03667417
Title: Genetic Predisposition to Breast and Ovarian Cancer: Prospective Study of BRCAx Gene Mutation
Acronym: GENEPSO
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: UNICANCER - Le Groupe génétique et cancer (GGC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: GENEPSO-IPC 2018-031
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancers; Ovarian Cancers
Keywords: BRCA gene mutation
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects carrying a BRCA gene mutation: subjects carrying a BRCA gene mutation
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — standardized data collection and 10-year prospective follow-up

SUMMARY:
Cohort of subjects carrying a BRCA gene mutation: genetic predispositions to breast and ovarian cancers

DETAILED DESCRIPTION:
Cohort of subjects carrying a BRCA gene mutation: genetic predispositions to breast and ovarian cancers

ELIGIBILITY:
1. Woman or man, with or without cancer, carrying a deleterious BRCA1/BRCA2 mutation, aged 18 years and over.

   1. Woman with or without breast cancer or ovarian cancer at baseline.
   2. Man with or without breast cancer at baseline.
2. Signed consent to participation
3. Affiliation to a social security regimen, or beneficiary of such a regimen.

Exclusion Criteria:

1. A person of legal age subject to a legal protection measure, or unable to express consent.
2. Impossibility to submit to the follow-up of the test for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women and men with a BRCA1 or BRCA2 mutation
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1999-10-15 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of breast and / or ovarian cancer during subject lifetime | 10 years
  risk that a subject with a mutation develops breast and / or ovarian cancer during his lifetime, assessed by epidemiologic questionnaires (carcinologic events).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine NOGUES, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pathology of familial breast cancer: differences between breast cancers in carriers of BRCA1 or BRCA2 mutations and sporadic cases. Breast Cancer Linkage Consortium. Lancet. 1997 May 24;349(9064):1505-10. PMID 9167459
- [Background] Brzovic PS, Meza J, King MC, Klevit RE. The cancer-predisposing mutation C61G disrupts homodimer formation in the NH2-terminal BRCA1 RING finger domain. J Biol Chem. 1998 Apr 3;273(14):7795-9. doi: 10.1074/jbc.273.14.7795. PMID 9525870
- [Background] Claus EB, Risch N, Thompson WD. Genetic analysis of breast cancer in the cancer and steroid hormone study. Am J Hum Genet. 1991 Feb;48(2):232-42. PMID 1990835
- [Background] Couch FJ, Weber BL. Mutations and polymorphisms in the familial early-onset breast cancer (BRCA1) gene. Breast Cancer Information Core. Hum Mutat. 1996;8(1):8-18. doi: 10.1002/humu.1380080102. PMID 8807330
- [Background] Den Otter W, Merchant TE, Beijerinck D, Koten JW. Breast cancer induction due to mammographic screening in hereditarily affected women. Anticancer Res. 1996 Sep-Oct;16(5B):3173-5. PMID 8967731
- [Background] Easton DF, Ford D, Bishop DT. Breast and ovarian cancer incidence in BRCA1-mutation carriers. Breast Cancer Linkage Consortium. Am J Hum Genet. 1995 Jan;56(1):265-71. PMID 7825587
- [Background] Easton D. Breast cancer genes--what are the real risks? Nat Genet. 1997 Jul;16(3):210-1. doi: 10.1038/ng0797-210. No abstract available. PMID 9207777
- [Background] Eisinger F, Thouvenin D, Bignon YJ, Cuisenier J, Feingold J, Hoerni B, Lasset C, Lyonnet D, Maraninchi D, Marty M, et al. [Considerations on the organization of oncologic-genetic consultations (a first step towards the publication of clinical practice guidelines)]. Bull Cancer. 1995 Oct;82(10):865-78. No abstract available. French. PMID 8535012
- [Background] Eisinger F, Stoppa-Lyonnet D, Longy M, Kerangueven F, Noguchi T, Bailly C, Vincent-Salomon A, Jacquemier J, Birnbaum D, Sobol H. Germ line mutation at BRCA1 affects the histoprognostic grade in hereditary breast cancer. Cancer Res. 1996 Feb 1;56(3):471-4. PMID 8564955
- [Background] Eisinger F, Jacquemier J, Charpin C, Stoppa-Lyonnet D, Bressac-de Paillerets B, Peyrat JP, Longy M, Guinebretiere JM, Sauvan R, Noguchi T, Birnbaum D, Sobol H. Mutations at BRCA1: the medullary breast carcinoma revisited. Cancer Res. 1998 Apr 15;58(8):1588-92. PMID 9563465
- [Background] Eisinger F, Alby N, Bremond A, Dauplat J, Espie M, Janiaud P, Kuttenn F, Lebrun JP, Lefranc JP, Pierret J, Sobol H, Stoppa-Lyonnet D, Thouvenin D, Tristant H, Feingold J. Recommendations for medical management of hereditary breast and ovarian cancer: the French National Ad Hoc Committee. Ann Oncol. 1998 Sep;9(9):939-50. doi: 10.1023/A:1008389021382. PMID 9818066
- [Background] Ford D, Easton DF, Bishop DT, Narod SA, Goldgar DE. Risks of cancer in BRCA1-mutation carriers. Breast Cancer Linkage Consortium. Lancet. 1994 Mar 19;343(8899):692-5. doi: 10.1016/s0140-6736(94)91578-4. PMID 7907678
- [Background] Ford D, Easton DF, Stratton M, Narod S, Goldgar D, Devilee P, Bishop DT, Weber B, Lenoir G, Chang-Claude J, Sobol H, Teare MD, Struewing J, Arason A, Scherneck S, Peto J, Rebbeck TR, Tonin P, Neuhausen S, Barkardottir R, Eyfjord J, Lynch H, Ponder BA, Gayther SA, Zelada-Hedman M, et al. Genetic heterogeneity and penetrance analysis of the BRCA1 and BRCA2 genes in breast cancer families. The Breast Cancer Linkage Consortium. Am J Hum Genet. 1998 Mar;62(3):676-89. doi: 10.1086/301749. PMID 9497246
- [Background] Gayther SA, Warren W, Mazoyer S, Russell PA, Harrington PA, Chiano M, Seal S, Hamoudi R, van Rensburg EJ, Dunning AM, Love R, Evans G, Easton D, Clayton D, Stratton MR, Ponder BA. Germline mutations of the BRCA1 gene in breast and ovarian cancer families provide evidence for a genotype-phenotype correlation. Nat Genet. 1995 Dec;11(4):428-33. doi: 10.1038/ng1295-428. PMID 7493024
- [Background] Gayther SA, Mangion J, Russell P, Seal S, Barfoot R, Ponder BA, Stratton MR, Easton D. Variation of risks of breast and ovarian cancer associated with different germline mutations of the BRCA2 gene. Nat Genet. 1997 Jan;15(1):103-5. doi: 10.1038/ng0197-103. PMID 8988179
- [Background] Hall JM, Lee MK, Newman B, Morrow JE, Anderson LA, Huey B, King MC. Linkage of early-onset familial breast cancer to chromosome 17q21. Science. 1990 Dec 21;250(4988):1684-9. doi: 10.1126/science.2270482.
- [Background] Houlston RS, Collins A, Slack J, Campbell S, Collins WP, Whitehead MI, Morton NE. Genetic epidemiology of ovarian cancer: segregation analysis. Ann Hum Genet. 1991 Oct;55(4):291-9. doi: 10.1111/j.1469-1809.1991.tb00856.x. PMID 1819229
- [Background] Julian-Reynier C, Eisinger F, Vennin P, Chabal F, Aurran Y, Nogues C, Bignon YJ, Machelard-Roumagnac M, Maugard-Louboutin C, Serin D, Blanc B, Orsoni P, Sobol H. Attitudes towards cancer predictive testing and transmission of information to the family. J Med Genet. 1996 Sep;33(9):731-6. doi: 10.1136/jmg.33.9.731. PMID 8880571
- [Background] Kerangueven F, Essioux L, Dib A, Noguchi T, Allione F, Geneix J, Longy M, Lidereau R, Eisinger F, Pebusque MJ, et al. Loss of heterozygosity and linkage analysis in breast carcinoma: indication for a putative third susceptibility gene on the short arm of chromosome 8. Oncogene. 1995 Mar 2;10(5):1023-6. PMID 7898921
- [Background] Lerman C, Narod S, Schulman K, Hughes C, Gomez-Caminero A, Bonney G, Gold K, Trock B, Main D, Lynch J, Fulmore C, Snyder C, Lemon SJ, Conway T, Tonin P, Lenoir G, Lynch H. BRCA1 testing in families with hereditary breast-ovarian cancer. A prospective study of patient decision making and outcomes. JAMA. 1996 Jun 26;275(24):1885-92. PMID 8648868
- [Background] Marcus JN, Watson P, Page DL, Narod SA, Lenoir GM, Tonin P, Linder-Stephenson L, Salerno G, Conway TA, Lynch HT. Hereditary breast cancer: pathobiology, prognosis, and BRCA1 and BRCA2 gene linkage. Cancer. 1996 Feb 15;77(4):697-709. doi: 10.1002/(sici)1097-0142(19960215)77:43.0.co;2-w. PMID 8616762
- [Background] Menegoz F, Black RJ, Arveux P, Magne V, Ferlay J, Buemi A, Carli PM, Chapelain G, Faivre J, Gignoux M, Grosclaude P, Mace-Lesec'h J, Raverdy N, Schaffer P. Cancer incidence and mortality in France in 1975-95. Eur J Cancer Prev. 1997 Oct;6(5):442-66. doi: 10.1097/00008469-199710000-00005. PMID 9466116
- [Background] Miki Y, Swensen J, Shattuck-Eidens D, Futreal PA, Harshman K, Tavtigian S, Liu Q, Cochran C, Bennett LM, Ding W, et al. A strong candidate for the breast and ovarian cancer susceptibility gene BRCA1. Science. 1994 Oct 7;266(5182):66-71. doi: 10.1126/science.7545954.
- [Background] Narod SA, Goldgar D, Cannon-Albright L, Weber B, Moslehi R, Ives E, Lenoir G, Lynch H. Risk modifiers in carriers of BRCA1 mutations. Int J Cancer. 1995 Dec 20;64(6):394-8. doi: 10.1002/ijc.2910640608. PMID 8550241
- [Background] Neuhausen SL, Mazoyer S, Friedman L, Stratton M, Offit K, Caligo A, Tomlinson G, Cannon-Albright L, Bishop T, Kelsell D, Solomon E, Weber B, Couch F, Struewing J, Tonin P, Durocher F, Narod S, Skolnick MH, Lenoir G, Serova O, Ponder B, Stoppa-Lyonnet D, Easton D, King MC, Goldgar DE. Haplotype and phenotype analysis of six recurrent BRCA1 mutations in 61 families: results of an international study. Am J Hum Genet. 1996 Feb;58(2):271-80. PMID 8571953
- [Background] NOGUES C et le groupe Génétique et Cancer de la FNCLCC (1996) Tests moléculaires dans le cancer du sein : attitude du Groupe Génétique et Cancer (GGC). Eurocancer 96, John Libbey Eurotext, Paris, pp. 177-178.
- [Background] Seitz S, Rohde K, Bender E, Nothnagel A, Kolble K, Schlag PM, Scherneck S. Strong indication for a breast cancer susceptibility gene on chromosome 8p12-p22: linkage analysis in German breast cancer families. Oncogene. 1997 Feb 13;14(6):741-3. doi: 10.1038/sj.onc.1200881. PMID 9038382
- [Background] Sobol H, Stoppa-Lyonnet D, Bressac-de-Paillerets B, Peyrat JP, Kerangueven F, Janin N, Noguchi T, Eisinger F, Guinebretiere JM, Jacquemier J, Birnbaum D. Truncation at conserved terminal regions of BRCA1 protein is associated with highly proliferating hereditary breast cancers. Cancer Res. 1996 Jul 15;56(14):3216-9. PMID 8764110
- [Background] Stoppa-Lyonnet D, Laurent-Puig P, Essioux L, Pages S, Ithier G, Ligot L, Fourquet A, Salmon RJ, Clough KB, Pouillart P, Bonaiti-Pellie C, Thomas G. BRCA1 sequence variations in 160 individuals referred to a breast/ovarian family cancer clinic. Institut Curie Breast Cancer Group. Am J Hum Genet. 1997 May;60(5):1021-30. PMID 9150149
- [Background] STOPPA-LYONNET D, NOGUES C, SOBOL H, EISINGER F (1998) Consultations de génétique et prédisposition au cancer du sein. In : Risques héréditaires de cancers du sein et de l'ovaire. Quelle prise en charge ? Expertise collective INSERM, Editions INSERM, Paris, pp. 179-189.
- [Background] Struewing JP, Hartge P, Wacholder S, Baker SM, Berlin M, McAdams M, Timmerman MM, Brody LC, Tucker MA. The risk of cancer associated with specific mutations of BRCA1 and BRCA2 among Ashkenazi Jews. N Engl J Med. 1997 May 15;336(20):1401-8. doi: 10.1056/NEJM199705153362001. PMID 9145676
- [Background] De VATHAIRE F, KOSCIELNY S, REZVANI A, LAPLANCHE A, ESTEVE J, FERLAY J (1996) Estimation de l'incidence des cancers en France 1983-1987. Editions INSERM, Paris.
- [Background] Verhoog LC, Brekelmans CT, Seynaeve C, van den Bosch LM, Dahmen G, van Geel AN, Tilanus-Linthorst MM, Bartels CC, Wagner A, van den Ouweland A, Devilee P, Meijers-Heijboer EJ, Klijn JG. Survival and tumour characteristics of breast-cancer patients with germline mutations of BRCA1. Lancet. 1998 Jan 31;351(9099):316-21. doi: 10.1016/s0140-6736(97)07065-7. PMID 9652611
- [Background] Wooster R, Neuhausen SL, Mangion J, Quirk Y, Ford D, Collins N, Nguyen K, Seal S, Tran T, Averill D, et al. Localization of a breast cancer susceptibility gene, BRCA2, to chromosome 13q12-13. Science. 1994 Sep 30;265(5181):2088-90. doi: 10.1126/science.8091231.
- [Background] Wooster R, Bignell G, Lancaster J, Swift S, Seal S, Mangion J, Collins N, Gregory S, Gumbs C, Micklem G. Identification of the breast cancer susceptibility gene BRCA2. Nature. 1995 Dec 21-28;378(6559):789-92. doi: 10.1038/378789a0. PMID 8524414
- [Result] Andrieu N, Easton DF, Chang-Claude J, Rookus MA, Brohet R, Cardis E, Antoniou AC, Wagner T, Simard J, Evans G, Peock S, Fricker JP, Nogues C, Van't Veer L, Van Leeuwen FE, Goldgar DE. Effect of chest X-rays on the risk of breast cancer among BRCA1/2 mutation carriers in the international BRCA1/2 carrier cohort study: a report from the EMBRACE, GENEPSO, GEO-HEBON, and IBCCS Collaborators' Group. J Clin Oncol. 2006 Jul 20;24(21):3361-6. doi: 10.1200/JCO.2005.03.3126. Epub 2006 Jun 26. PMID 16801631
- [Result] Lecarpentier J, Nogues C, Mouret-Fourme E, Gauthier-Villars M, Lasset C, Fricker JP, Caron O, Stoppa-Lyonnet D, Berthet P, Faivre L, Bonadona V, Buecher B, Coupier I, Gladieff L, Gesta P, Eisinger F, Frenay M, Luporsi E, Lortholary A, Colas C, Dugast C, Longy M, Pujol P, Tinat J; GENEPSO; Lidereau R, Andrieu N. Variation in breast cancer risk associated with factors related to pregnancies according to truncating mutation location, in the French National BRCA1 and BRCA2 mutations carrier cohort (GENEPSO). Breast Cancer Res. 2012 Jul 3;14(4):R99. doi: 10.1186/bcr3218. PMID 22762150
- [Result] GENEPSO : cohorte nationale prospective de personnes porteuses d'une mutation sur les gènes BRCA1 et BRCA2 GENEPSO: French BRCA1/2 carrier cohort study E. Fourme, C. Picard, M.L. Manche-Thévenot, C. Noguès, groupe Génétique et cancer* La Lettre du Sénologue • n° 43 - janvier-février-mars 2009
- [Result] Bonaiti B, Alarcon F, Bonadona V, Pennec S, Andrieu N, Stoppa-Lyonnet D, Perdry H, Bonaiti-Pellie C; Groupe Genetique et Cancer. [A new scoring system for the diagnosis of BRCA1/2 associated breast-ovarian cancer predisposition]. Bull Cancer. 2011 Jul;98(7):779-95. doi: 10.1684/bdc.2011.1397. French. PMID 21708517
- [Result] Eisinger F, Bressac B, Castaigne D, Cottu PH, Lansac J, Lefranc JP, Lesur A, Nogues C, Pierret J, Puy-Pernias S, Sobol H, Tardivon A, Tristant H, Villet R. [Identification and management of hereditary predisposition to cancer of the breast and the ovary (update 2004)]. Bull Cancer. 2004 Mar;91(3):219-37. French. PMID 15171047
- [Result] Kuchenbaecker KB, Hopper JL, Barnes DR, Phillips KA, Mooij TM, Roos-Blom MJ, Jervis S, van Leeuwen FE, Milne RL, Andrieu N, Goldgar DE, Terry MB, Rookus MA, Easton DF, Antoniou AC; BRCA1 and BRCA2 Cohort Consortium; McGuffog L, Evans DG, Barrowdale D, Frost D, Adlard J, Ong KR, Izatt L, Tischkowitz M, Eeles R, Davidson R, Hodgson S, Ellis S, Nogues C, Lasset C, Stoppa-Lyonnet D, Fricker JP, Faivre L, Berthet P, Hooning MJ, van der Kolk LE, Kets CM, Adank MA, John EM, Chung WK, Andrulis IL, Southey M, Daly MB, Buys SS, Osorio A, Engel C, Kast K, Schmutzler RK, Caldes T, Jakubowska A, Simard J, Friedlander ML, McLachlan SA, Machackova E, Foretova L, Tan YY, Singer CF, Olah E, Gerdes AM, Arver B, Olsson H. Risks of Breast, Ovarian, and Contralateral Breast Cancer for BRCA1 and BRCA2 Mutation Carriers. JAMA. 2017 Jun 20;317(23):2402-2416. doi: 10.1001/jama.2017.7112. PMID 28632866
- [Result] Mancini J, Le Cozannet E, Bouhnik AD, Resseguier N, Lasset C, Mouret-Fourme E, Nogues C, Julian-Reynier C. Disclosure of research results: a randomized study on GENEPSO-PS cohort participants. Health Expect. 2016 Oct;19(5):1023-35. doi: 10.1111/hex.12390. Epub 2015 Jul 23. PMID 26205609
- [Result] Lecarpentier J, Nogues C, Mouret-Fourme E, Buecher B, Gauthier-Villars M, Stoppa-Lyonnet D, Bonadona V, Fricker JP, Berthet P, Caron O, Coupier I, Pujol P, Faivre L, Gesta P, Eisinger F, Mari V, Gladieff L, Lortholary A, Luporsi E, Leroux D, Venat-Bouvet L, Maugard CM, Colas C, Tinat J, Lasset C, Andrieu N; GENEPSO. Breast Cancer Risk Associated with Estrogen Exposure and Truncating Mutation Location in BRCA1/2 Carriers. Cancer Epidemiol Biomarkers Prev. 2015 Apr;24(4):698-707. doi: 10.1158/1055-9965.EPI-14-0884. Epub 2015 Jan 22. PMID 25613119
- [Result] Julian-Reynier C, Resseguier N, Bouhnik AD, Eisinger F, Lasset C, Fourme E, Nogues C. Cigarette smoking in women after BRCA1/2 genetic test disclosure: a 5-year follow-up study of the GENEPSO PS cohort. Genet Med. 2015 Feb;17(2):117-24. doi: 10.1038/gim.2014.82. Epub 2014 Jul 10. PMID 25010056
- [Result] Bureau E, Pellegrini I, Nogues C, Lasset C, Julian-Reynier C. "Maybe they have found something new" participants' views on returning cohort psychosocial survey results. Health Expect. 2015 Dec;18(6):2425-36. doi: 10.1111/hex.12211. Epub 2014 May 30. PMID 24889689
- [Result] Lapointe J, Dorval M, Nogues C, Fabre R; GENEPSO Cohort; Julian-Reynier C. Is the psychological impact of genetic testing moderated by support and sharing of test results to family and friends? Fam Cancer. 2013 Dec;12(4):601-10. doi: 10.1007/s10689-013-9621-3. PMID 23475556
- [Result] Pijpe A, Andrieu N, Easton DF, Kesminiene A, Cardis E, Nogues C, Gauthier-Villars M, Lasset C, Fricker JP, Peock S, Frost D, Evans DG, Eeles RA, Paterson J, Manders P, van Asperen CJ, Ausems MG, Meijers-Heijboer H, Thierry-Chef I, Hauptmann M, Goldgar D, Rookus MA, van Leeuwen FE; GENEPSO; EMBRACE; HEBON. Exposure to diagnostic radiation and risk of breast cancer among carriers of BRCA1/2 mutations: retrospective cohort study (GENE-RAD-RISK). BMJ. 2012 Sep 6;345:e5660. doi: 10.1136/bmj.e5660. PMID 22956590
- [Result] Eisinger F, Fabre R, Lasset C, Stoppa-Lyonnet D, Julian-Reynier C, Nogues C. Spontaneous disclosure of BRCA1/2 genetic test results to employers: a French prospective study. Eur J Hum Genet. 2012 Sep;20(9):981-3. doi: 10.1038/ejhg.2012.37. Epub 2012 Feb 29. PMID 22378286
- [Result] Pujol P, Lasset C, Berthet P, Dugast C, Delaloge S, Fricker JP, Tennevet I, Chabbert-Buffet N, This P, Baudry K, Lemonnier J, Roca L, Mijonnet S, Gesta P, Chiesa J, Dreyfus H, Vennin P, Delnatte C, Bignon YJ, Lortholary A, Prieur F, Gladieff L, Lesur A, Clough KB, Nogues C, Martin AL; French Federation of Cancer Centres (FNCLCC). Uptake of a randomized breast cancer prevention trial comparing letrozole to placebo in BRCA1/2 mutations carriers: the LIBER trial. Fam Cancer. 2012 Mar;11(1):77-84. doi: 10.1007/s10689-011-9484-4. PMID 22076253
- [Result] Lecarpentier J, Nogues C, Mouret-Fourme E, Stoppa-Lyonnet D, Lasset C, Caron O, Fricker JP, Gladieff L, Faivre L, Sobol H, Gesta P, Frenay M, Luporsi E, Coupier I; GENEPSO; Lidereau R, Andrieu N. Variation in breast cancer risk with mutation position, smoking, alcohol, and chest X-ray history, in the French National BRCA1/2 carrier cohort (GENEPSO). Breast Cancer Res Treat. 2011 Dec;130(3):927-38. doi: 10.1007/s10549-011-1655-3. Epub 2011 Jul 15. PMID 21761160
- [Result] Dorval M, Nogues C, Berthet P, Chiquette J, Gauthier-Villars M, Lasset C, Picard C, Plante M; INHERIT BRCAs; GENEPSO Cohort; Simard J, Julian-Reynier C. Breast and ovarian cancer screening of non-carriers from BRCA1/2 mutation-positive families: 2-year follow-up of cohorts from France and Quebec. Eur J Hum Genet. 2011 May;19(5):494-9. doi: 10.1038/ejhg.2010.227. Epub 2011 Jan 19. PMID 21248744
- [Result] Antoniou AC, Rookus M, Andrieu N, Brohet R, Chang-Claude J, Peock S, Cook M, Evans DG, Eeles R; EMBRACE; Nogues C, Faivre L, Gesta P; GENEPSO; van Leeuwen FE, Ausems MG, Osorio A; GEO-HEBON; Caldes T, Simard J, Lubinski J, Gerdes AM, Olah E, Furhauser C, Olsson H, Arver B, Radice P, Easton DF, Goldgar DE. Reproductive and hormonal factors, and ovarian cancer risk for BRCA1 and BRCA2 mutation carriers: results from the International BRCA1/2 Carrier Cohort Study. Cancer Epidemiol Biomarkers Prev. 2009 Feb;18(2):601-10. doi: 10.1158/1055-9965.EPI-08-0546. Epub 2009 Feb 3. PMID 19190154
- [Result] Brohet RM, Goldgar DE, Easton DF, Antoniou AC, Andrieu N, Chang-Claude J, Peock S, Eeles RA, Cook M, Chu C, Nogues C, Lasset C, Berthet P, Meijers-Heijboer H, Gerdes AM, Olsson H, Caldes T, van Leeuwen FE, Rookus MA. Oral contraceptives and breast cancer risk in the international BRCA1/2 carrier cohort study: a report from EMBRACE, GENEPSO, GEO-HEBON, and the IBCCS Collaborating Group. J Clin Oncol. 2007 Sep 1;25(25):3831-6. doi: 10.1200/JCO.2007.11.1179. Epub 2007 Jul 16. PMID 17635951
- [Result] Chang-Claude J, Andrieu N, Rookus M, Brohet R, Antoniou AC, Peock S, Davidson R, Izatt L, Cole T, Nogues C, Luporsi E, Huiart L, Hoogerbrugge N, Van Leeuwen FE, Osorio A, Eyfjord J, Radice P, Goldgar DE, Easton DF; Epidemiological Study of Familial Breast Cancer (EMBRACE); Gene Etude Prospective Sein Ovaire (GENEPSO); Genen Omgeving studie van de werkgroep Hereditiair Borstkanker Onderzoek Nederland (GEO-HEBON); International BRCA1/2 Carrier Cohort Study (IBCCS) collaborators group. Age at menarche and menopause and breast cancer risk in the International BRCA1/2 Carrier Cohort Study. Cancer Epidemiol Biomarkers Prev. 2007 Apr;16(4):740-6. doi: 10.1158/1055-9965.EPI-06-0829. PMID 17416765
- [Result] Andrieu N, Goldgar DE, Easton DF, Rookus M, Brohet R, Antoniou AC, Peock S, Evans G, Eccles D, Douglas F, Nogues C, Gauthier-Villars M, Chompret A, Van Leeuwen FE, Kluijt I, Benitez J, Arver B, Olah E, Chang-Claude J; EMBRACE; GENEPSO; GEO-HEBON; IBCCS Collaborators Group. Pregnancies, breast-feeding, and breast cancer risk in the International BRCA1/2 Carrier Cohort Study (IBCCS). J Natl Cancer Inst. 2006 Apr 19;98(8):535-44. doi: 10.1093/jnci/djj132. PMID 16622123
- [Result] Jegu M, Some Der A, Morcel K, Abadie C, Fritel X, Leveque J. [Breast and ovarian cancer due to BRCA1&2 hereditary cancer predisposition syndrome and reproduction: literature review]. J Gynecol Obstet Biol Reprod (Paris). 2015 Jan;44(1):10-7. doi: 10.1016/j.jgyn.2014.10.011. Epub 2014 Nov 18. French. PMID 25455630
- [Result] Feunteun J. [A paradox and three egnimas about the role of BRCA1 in breast and ovarian cancers]. J Soc Biol. 2004;198(2):123-6. French. PMID 15368961
- [Result] Suivi prospectif à 5 ans des tests de prédisposition génétique au cancer du sein et/ou de l'ovaire : comportements de prévention, attentes envers la recherche et inégalités sociales (cohorte nationale Genepso) Institut National du Cancer (INCa) dans le cadre de l'appel à projets 2011 Projets libres de recherché en sciences humaines et sociales, épidémiologie et santé publique.
- [Result] Bonaiti-Pellie C, Andrieu N, Arveux P, Bonadona V, Buecher B, Delpech M, Jolly D, Julian-Reynier C, Luporsi E, Nogues C, Nowak F, Olschwang S, Orsi F, Pujol P, Saurin JC, Sinilnikova O, Stoppa-Lyonnet D, Thepot F. [Cancer genetics: estimation of the needs of the population in France for the next ten years]. Bull Cancer. 2009 Sep;96(9):875-900. doi: 10.1684/bdc.2009.0943. French. PMID 19751997
- See also: Description de la cohorte GENEPSO au sein du Portail Epidémiologie-France — https://epidemiologie-france.aviesan.fr/epidemiologie-france/fiches/cohorte-de-sujets-portant-une-mutation-des-genes-brca-predispositions-genetiques-aux-cancers-du-sein-et-de-l-ovaire/fre-fr